CLINICAL TRIAL: NCT06289673
Title: INITIALL: Identification of Necessary Information for Treatment Induction in Newly Diagnosed Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: Identification of Necessary Information for Treatment Induction in Newly Diagnosed Acute Lymphoblastic Leukemia/Lymphoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INITIALL; NCI-2024-01659 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-02-23; First posted 2024-03-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Mixed Phenotype Acute Leukemia
Keywords: Newly Diagnosed; Risk Category; Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Mixed Phenotype Acute Leukemia (MPAL); Children; Young Adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — Dexamethasone; Calcium Dobesilate; Vincristine; Daunorubicin; Methotrexate; Hydrocortisone; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Newly diagnosed ALL, LLy, and MPAL patients (Experimental): All eligible patients receive the following intervention:
  Dexamethasone, Vincristine, Daunorubicin, Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine)
  Interventions: Drug: Dexamethasone; Drug: Vincristine; Drug: Daunorubicin; Drug: Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine); Drug: Methotrexate; Drug: Cytarabine

INTERVENTIONS:
Drug: Dexamethasone — Per mouth (PO) or intravenously (IV) once on Day 1 and PO or IV divided BID (every 12 hours) days 2-7
  Other Names: Decadron
Drug: Vincristine — Intravenously (IV) for 1 dose on Day 1 or 2
  Other Names: Vincristine Sulfate; Oncovin
Drug: Daunorubicin — Intravenously (IV) for 1 dose on Day 2 or 3 (T-ALL/ T-LLy/ MPAL only)
  Other Names: Daunomycin
Drug: Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine) — Intrathecal (Age adjusted) for 1 dose on Day 4 or 5 or 6
  Other Names: ITMHA
Drug: Methotrexate — Given IT as part of Intrathecal triple therapy.
  Other Names: MTX; Trexall®
Drug: Cytarabine — Given IT as part of Intrathecal triple therapy.
  Other Names: Cytosine arabinoside; Ara-C

SUMMARY:
The goal of this study is to provide sufficient therapy during the time a patients' B-cell Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LLy) risk category is being determined. The term "risk" refers to the chance of the ALL or LLy coming back after treatment.

Primary Objectives

* To provide sufficient therapy to enable testing of newly diagnosed acute lymphoblastic leukemia/lymphoma and mixed phenotype acute leukemia/lymphoma tumor samples to determine eligibility and appropriate risk stratification for SJALL therapeutic studies.
* To develop a central database of genomic and clinical findings.

Secondary Objectives

* To assess event free and overall survival data of patients enrolled on this study.

DETAILED DESCRIPTION:
Patients with newly diagnosed acute lymphoblastic leukemia/lymphoma (ALL/LLy) and mixed phenotype acute leukemia/lymphoma (MPAL) will undergo diagnostic procedures either during screening or on Day 1. They will receive 7 days of chemotherapy including 13 doses of dexamethasone, 1 dose of vincristine, and 1 dose of daunorubicin (for patients with T-ALL/LLy or MPAL only). Patients will also undergo their initial lumbar puncture with intrathecal chemotherapy on Days 4 or 5 or 6 of therapy. After the completion of 7 days of chemotherapy, patients will begin therapy on either a SJALL therapeutic trial or will receive non-protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-18.99 years
* Diagnosis of acute leukemia / lymphoma as below:

  * Acute lymphoblastic leukemia (ALL) with at least 25% bone marrow blasts or definitive evidence of ALL in peripheral blood (in those without an available bone marrow sample).
  * Lymphoblastic lymphoma (LLy) with immunophenotypic evidence of a lymphoblastic population and <25% bone marrow blasts and less than 1,000 circulating blasts/ microL.
  * Mixed phenotype acute leukemia (MPAL) with or without 25% bone marrow involvement (i.e. patients with either leukemia or lymphoma are eligible).

Exclusion Criteria:

* Pregnant or breastfeeding
* Receipt of prior cancer directed therapy with the exclusion of up to 1 dose of intrathecal chemotherapy, 1 dose of vincristine, or emergency radiotherapy due to organ compromising malignant mass. There is no exclusion for prior steroid therapy.
* Known to be currently ineligible for available SJALL therapeutic studies (e.g. receipt of prohibited therapy, no appropriate SJALL therapeutic study available, enrolled on competing trial, etc.).

Note: The intention of this exclusion criterion is to enroll all newly diagnosed ALL/ LLy/ MPAL patients. If participant is screened as a potential participant for subsequent SJALL and later found to be ineligible due to information obtained during INITIALL, this will not make the participant ineligible for INITIALL.

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Major pre-existing abnormalities such as ataxia telangiectasia, Fanconi anemia, Charcot Marie Tooth, etc.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 850 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2034-05 (Estimated); Study Completion 2039-05 (Estimated)

PRIMARY OUTCOMES:
Sufficient phenotypic and/or genomic data necessary for therapeutic protocol assignment by Day 8 (completion of INITIALL therapy). | 1 week from study entry
  The proportion of patients with sufficient immunophenotypic, genomic, and clinical data to allow determination of eligibility for currently open trials at the enrolling institution.
Complete data within the INITIALL database | 3 months, 1 year, 3, 5 years from study entry
  The proportion of patients with complete data within the INITIALL protocol database as described in the protocol.

SECONDARY OUTCOMES:
Event Free Survival (EFS) | 1, 3, 5 years from study entry
  EFS will be reported as estimates using the Kaplan-Meier method.
Overall Survival (OS) | 1, 3, 5 years from study entry
  OS will be reported as estimates using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Seth E. Karol, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Rady Children's Hospital, San Diego, California
  - Saint Francis Children's Hospital, Tulsa, Oklahoma
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols